CLINICAL TRIAL: NCT03713333
Title: Implementation of High Definition Screening Using Handheld Imaging and Digital Health Technologies Within a Learning Health System to Identify Cardiovascular Disease at the Point-of-care: The ASE-INNOVATE Program
Brief Title: Implementing Digital Health in a Learning Health System
Acronym: ASE-INNOVATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Health (Other)
Collaborators: West Virginia University (Other)
Responsible Party: Principal Investigator, Sanjeev Bhavnani MD, Principal Investigator - Healthcare Innovation, Scripps Health
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Screening
Other Study IDs: Pro00029622
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Cardiovascular Diseases; Hypertension; Heart Failure; Atrial Fibrillation; Metabolic Syndrome; Genetic Disease
Keywords: digital health; handheld ultrasound; smartphone ECG; mobile health; point of care genomics; big data; artificial intelligence; learning health system
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Heart Failure; Atrial Fibrillation; Metabolic Syndrome; Genetic Diseases, Inborn

STUDY DESIGN:
Intervention Model Description: Pragmatic, multisite, cluster randomized trial comparing point of care and remote patient monitoring with digital health devices and handheld imaging to standard-care
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Treating physicians and clinical practitioners will not be concealed to the randomized allocation of individual clinics or the patients that are seen in these encounters. Physicians in the interventional group will participate in conducting technology-enabled visitations before and after a patient encounter and therefore are not blinded to the assessment. For the standard care group handheld imaging and remote patient monitoring will not be performed after the patient-physician encounter. Principal investigators, outcome adjudicators, and statisticians are blinded to randomization, device findings, and treatment decisions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Technology-Enabled Visitations (Experimental): Technology-enabled visitations with digital health will include the following devices used at the time of a patient-physician encounter. These findings will be available to the treating physician at the time the visitation and to be used for clinical decisions.
  Interventions: Diagnostic Test: Digital Health Device Diagnostics
- Standard-Care Visitations (No Intervention): Standard-care is defined as the range of services available during usual patient care. Handheld Imaging and digital health screening will be performed in the control group after the patient-physician encounter. As such, patients and physicians will be blinded to the diagnostic findings unless an abnormal finding is detected that requires physician review and triage for further care.

INTERVENTIONS:
Diagnostic Test: Digital Health Device Diagnostics — Technology-enabled visitations with digital health will include the following devices used at the time of a patient-physician encounter. These findings will be available to the treating physician at the time the visitation and to be used for clinical decisions.
  * Handheld imaging - focused echocardiographic examination (Butterfly IQ)
  * Smartphone iECG for cardiac rhythm assessments (Alivecor)
  * Blood Pressure (CloudDX)
  * Oxygen Saturation (CloudDX)
  * Weight (CloudDX)
  * Point-of-Care Genetic Testing (Phosphorous)
  Arms: Technology-Enabled Visitations

SUMMARY:
The need for new models of integrated care that can improve the efficiency of healthcare and reduce the costs are key priorities for health systems across the United States. Treatment costs for patients with at least one chronic medical or cardiovascular condition make up over 4-trillion dollars in spending on healthcare, with estimations of a population prevalence of 100-million affected individuals within the next decade. Therefore, the management of chronic conditions requires innovative and new implementation methods that improve outcomes, reduce costs, and increase healthcare efficiencies. Digital health, the use of mobile computing and communication technologies as an integral new models of care is seen as one potential solution. Despite the potential applications, there is limited data to support that new technologies improve healthcare outcomes. To do so requires; 1) robust methods to determine the impact of new technologies on healthcare outcomes and costs; and 2) evaluative mechanisms for how new devices are integrated into patient care. In this regard, the proposed clinical trial aims to advance the investigator's knowledge and to demonstrate the pragmatic utilization of new technologies within a learning healthcare system providing services to high-risk patient populations.

DETAILED DESCRIPTION:
Objective #1: Determine the effectiveness of handheld imaging and digital health devices on long term health and patient-reported outcomes through pragmatic and randomized clinical trial designs.

Objective #2: Assess the impact of digital health devices and remote patient monitoring (RPM) on measures of healthcare efficiency. Measures of healthcare efficiency directly related to digital health technologies and RPM include: identify which interventions can improve care; define the variations in care and; demonstrate within which patient populations digital health technologies are most effective.

Objective #3: Apply integration methods for handheld imaging and digital health devices used for clinical decisions.

Achieving integration and interoperability-the ability of different information technology systems and software applications to communicate and exchange data with each other-requires identiﬁcation for precisely how new innovations merge into systems of care and are applied to various practice settings.

ELIGIBILITY:
Inclusion Criteria:

* All participants of the ASE 2018 Outreach Event who are at least 18 years old who are referred for a cardiac evaluation

Exclusion Criteria:

* Those not willing to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2018-10-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Health Economic Outcomes | 180 days
  Economic difference between the total costs of care between randomized arms including; clinic visitations, hospitalizations, emergency room visitations, and diagnostic testing. Collected as cumulative diagnosis-related group (DRG) and current procedural terminology (CPT) amounts in United States Dollars

SECONDARY OUTCOMES:
Mobile Cardiac Telemetry | 180 days
  Number of referrals for mobile cardiac telemetry monitoring between randomized arms
Health Economic Outcomes | 30 days
  Economic difference between the total costs of care between randomized arms including; clinic visitations, hospitalizations, emergency room visitations, and diagnostic testing. Collected as cumulative diagnosis-related group (DRG) and current procedural terminology (CPT) amounts in United States Dollars
Patient-Reported Outcome Measures | 30 days
  Veterans Research and Development Corporation-12 Patient Reported Outcomes (mean total score 50 +/- 10) where higher values are associated with greater mental and physical debility
Patient-Reported Outcome Measures | 180 days
  Veterans Research and Development Corporation-12 Patient Reported Outcomes (mean total score 50 +/- 10) where higher values are associated with greater mental and physical debility
Patient-Reported Experience Measures | 30 days
  Agency for Healthcare Research and Quality Consumer Assessment of Healthcare Providers and Systems (average scores and difference between randomized arms) where higher scores are associated with greater patient satisfaction and patient experience
Patient-Reported Experience Measures | 180 days
  Agency for Healthcare Research and Quality Consumer Assessment of Healthcare Providers and Systems (average scores and difference between randomized arms) where higher scores are associated with greater patient satisfaction and patient experience
Diagnostic Imaging | 180 days
  Number of referrals for diagnostic imaging with transthoracic echocardiography between randomized arms
Heart Failure | 180 days
  Incidence of heart failure diagnosed between randomized arms
Atrial Fibrillation | 180 days
  Incidence of atrial fibrillation diagnosed between randomized arms
Emergency Department Visitations | 180 days
  Percentage of patients presenting to the emergency department for a cardiac condition (example; myocardial infarction, heart failure, atrial fibrillation, and stroke) between randomized arms
Hospitalization | 180 days
  Percentage of patients hospitalized for a cardiac condition (example; myocardial infarction, heart failure, atrial fibrillation, and stroke) between randomized arms
Clinic Visitations | 180 days
  Percentage of patients presenting for a clinical visitation for a cardiac condition (example; myocardial infarction, heart failure, atrial fibrillation, and stroke) between randomized arms
Medical Therapy | 180 days
  Percentage of patients initiating medical therapy for a cardiac condition including: heart failure, coronary artery disease, atrial fibrillation, and/or hypertension between randomized arms

CONTACTS AND LOCATIONS:
Overall Officials: Partho Sengupta, MD, Principal Investigator — West Virginia University Heart and Vascular Institute; Sanjeev Bhavnani, MD, Study Director — Scripps Clinic
Locations (1):
- West Virgina University, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singh S, Bansal M, Maheshwari P, Adams D, Sengupta SP, Price R, Dantin L, Smith M, Kasliwal RR, Pellikka PA, Thomas JD, Narula J, Sengupta PP; ASE-REWARD Study Investigators. American Society of Echocardiography: Remote Echocardiography with Web-Based Assessments for Referrals at a Distance (ASE-REWARD) Study. J Am Soc Echocardiogr. 2013 Mar;26(3):221-33. doi: 10.1016/j.echo.2012.12.012. PMID 23439071
- [Background] Bansal M, Sengupta PP. How to interpret an echocardiography report (for the non-imager)? Heart. 2017 Nov;103(21):1733-1744. doi: 10.1136/heartjnl-2016-309443. Epub 2017 Sep 7. No abstract available. PMID 28883036
- [Background] Bansal M, Sengupta PP. Setting global standards in adult echocardiography: Where are we? Indian Heart J. 2015 Jul-Aug;67(4):298-301. doi: 10.1016/j.ihj.2015.07.020. Epub 2015 Aug 21. No abstract available. PMID 26304560
- [Background] Bhavnani SP, Parakh K, Atreja A, Druz R, Graham GN, Hayek SS, Krumholz HM, Maddox TM, Majmudar MD, Rumsfeld JS, Shah BR. 2017 Roadmap for Innovation-ACC Health Policy Statement on Healthcare Transformation in the Era of Digital Health, Big Data, and Precision Health: A Report of the American College of Cardiology Task Force on Health Policy Statements and Systems of Care. J Am Coll Cardiol. 2017 Nov 28;70(21):2696-2718. doi: 10.1016/j.jacc.2017.10.018. No abstract available. PMID 29169478
- [Background] Chamsi-Pasha MA, Sengupta PP, Zoghbi WA. Handheld Echocardiography: Current State and Future Perspectives. Circulation. 2017 Nov 28;136(22):2178-2188. doi: 10.1161/CIRCULATIONAHA.117.026622. PMID 29180495
- [Background] Levine DM, Linder JA, Landon BE. The Quality of Outpatient Care Delivered to Adults in the United States, 2002 to 2013. JAMA Intern Med. 2016 Dec 1;176(12):1778-1790. doi: 10.1001/jamainternmed.2016.6217. PMID 27749962
- [Background] Maddox TM, Albert NM, Borden WB, Curtis LH, Ferguson TB Jr, Kao DP, Marcus GM, Peterson ED, Redberg R, Rumsfeld JS, Shah ND, Tcheng JE; American Heart Association Council on Quality of Care and Outcomes Research; Council on Cardiovascular Disease in the Young; Council on Clinical Cardiology; Council on Functional Genomics and Translational Biology; and Stroke Council. The Learning Healthcare System and Cardiovascular Care: A Scientific Statement From the American Heart Association. Circulation. 2017 Apr 4;135(14):e826-e857. doi: 10.1161/CIR.0000000000000480. Epub 2017 Mar 2. PMID 28254835
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Henderson C, Knapp M, Fernandez JL, Beecham J, Hirani SP, Beynon M, Cartwright M, Rixon L, Doll H, Bower P, Steventon A, Rogers A, Fitzpatrick R, Barlow J, Bardsley M, Newman SP. Cost-effectiveness of telecare for people with social care needs: the Whole Systems Demonstrator cluster randomised trial. Age Ageing. 2014 Nov;43(6):794-800. doi: 10.1093/ageing/afu067. Epub 2014 Jun 20. PMID 24950690
- [Background] Delaney SK, Hultner ML, Jacob HJ, Ledbetter DH, McCarthy JJ, Ball M, Beckman KB, Belmont JW, Bloss CS, Christman MF, Cosgrove A, Damiani SA, Danis T, Delledonne M, Dougherty MJ, Dudley JT, Faucett WA, Friedman JR, Haase DH, Hays TS, Heilsberg S, Huber J, Kaminsky L, Ledbetter N, Lee WH, Levin E, Libiger O, Linderman M, Love RL, Magnus DC, Martland A, McClure SL, Megill SE, Messier H, Nussbaum RL, Palaniappan L, Patay BA, Popovich BW, Quackenbush J, Savant MJ, Su MM, Terry SF, Tucker S, Wong WT, Green RC. Toward clinical genomics in everyday medicine: perspectives and recommendations. Expert Rev Mol Diagn. 2016;16(5):521-32. doi: 10.1586/14737159.2016.1146593. Epub 2016 Feb 24. PMID 26810587
- [Background] Orlando LA, Sperber NR, Voils C, Nichols M, Myers RA, Wu RR, Rakhra-Burris T, Levy KD, Levy M, Pollin TI, Guan Y, Horowitz CR, Ramos M, Kimmel SE, McDonough CW, Madden EB, Damschroder LJ. Developing a common framework for evaluating the implementation of genomic medicine interventions in clinical care: the IGNITE Network's Common Measures Working Group. Genet Med. 2018 Jun;20(6):655-663. doi: 10.1038/gim.2017.144. Epub 2017 Sep 14. PMID 28914267
- [Background] Via G, Hussain A, Wells M, Reardon R, ElBarbary M, Noble VE, Tsung JW, Neskovic AN, Price S, Oren-Grinberg A, Liteplo A, Cordioli R, Naqvi N, Rola P, Poelaert J, Gulic TG, Sloth E, Labovitz A, Kimura B, Breitkreutz R, Masani N, Bowra J, Talmor D, Guarracino F, Goudie A, Xiaoting W, Chawla R, Galderisi M, Blaivas M, Petrovic T, Storti E, Neri L, Melniker L; International Liaison Committee on Focused Cardiac UltraSound (ILC-FoCUS); International Conference on Focused Cardiac UltraSound (IC-FoCUS). International evidence-based recommendations for focused cardiac ultrasound. J Am Soc Echocardiogr. 2014 Jul;27(7):683.e1-683.e33. doi: 10.1016/j.echo.2014.05.001. PMID 24951446
- [Background] Spencer KT, Kimura BJ, Korcarz CE, Pellikka PA, Rahko PS, Siegel RJ. Focused cardiac ultrasound: recommendations from the American Society of Echocardiography. J Am Soc Echocardiogr. 2013 Jun;26(6):567-81. doi: 10.1016/j.echo.2013.04.001. No abstract available. PMID 23711341
- [Result] Bhavnani SP, Sola S, Adams D, Venkateshvaran A, Dash PK, Sengupta PP; ASEF-VALUES Investigators. A Randomized Trial of Pocket-Echocardiography Integrated Mobile Health Device Assessments in Modern Structural Heart Disease Clinics. JACC Cardiovasc Imaging. 2018 Apr;11(4):546-557. doi: 10.1016/j.jcmg.2017.06.019. Epub 2017 Oct 5. PMID 28917688
- [Result] Bhavnani SP, Narula J, Sengupta PP. Mobile technology and the digitization of healthcare. Eur Heart J. 2016 May 7;37(18):1428-38. doi: 10.1093/eurheartj/ehv770. Epub 2016 Feb 11. PMID 26873093
- [Result] Bansal M, Singh S, Maheshwari P, Adams D, McCulloch ML, Dada T, Sengupta SP, Kasliwal RR, Pellikka PA, Sengupta PP; VISION-in-Tele-Echo Study Investigators. Value of interactive scanning for improving the outcome of new-learners in transcontinental tele-echocardiography (VISION-in-Tele-Echo) study. J Am Soc Echocardiogr. 2015 Jan;28(1):75-87. doi: 10.1016/j.echo.2014.09.001. Epub 2014 Oct 8. PMID 25306222
- [Result] Lowres N, Neubeck L, Salkeld G, Krass I, McLachlan AJ, Redfern J, Bennett AA, Briffa T, Bauman A, Martinez C, Wallenhorst C, Lau JK, Brieger DB, Sy RW, Freedman SB. Feasibility and cost-effectiveness of stroke prevention through community screening for atrial fibrillation using iPhone ECG in pharmacies. The SEARCH-AF study. Thromb Haemost. 2014 Jun;111(6):1167-76. doi: 10.1160/TH14-03-0231. Epub 2014 Apr 1. PMID 24687081
- [Result] Kaczorowski J, Chambers LW, Dolovich L, Paterson JM, Karwalajtys T, Gierman T, Farrell B, McDonough B, Thabane L, Tu K, Zagorski B, Goeree R, Levitt CA, Hogg W, Laryea S, Carter MA, Cross D, Sabaldt RJ. Improving cardiovascular health at population level: 39 community cluster randomised trial of Cardiovascular Health Awareness Program (CHAP). BMJ. 2011 Feb 7;342:d442. doi: 10.1136/bmj.d442. PMID 21300712
- [Result] US Burden of Disease Collaborators; Mokdad AH, Ballestros K, Echko M, Glenn S, Olsen HE, Mullany E, Lee A, Khan AR, Ahmadi A, Ferrari AJ, Kasaeian A, Werdecker A, Carter A, Zipkin B, Sartorius B, Serdar B, Sykes BL, Troeger C, Fitzmaurice C, Rehm CD, Santomauro D, Kim D, Colombara D, Schwebel DC, Tsoi D, Kolte D, Nsoesie E, Nichols E, Oren E, Charlson FJ, Patton GC, Roth GA, Hosgood HD, Whiteford HA, Kyu H, Erskine HE, Huang H, Martopullo I, Singh JA, Nachega JB, Sanabria JR, Abbas K, Ong K, Tabb K, Krohn KJ, Cornaby L, Degenhardt L, Moses M, Farvid M, Griswold M, Criqui M, Bell M, Nguyen M, Wallin M, Mirarefin M, Qorbani M, Younis M, Fullman N, Liu P, Briant P, Gona P, Havmoller R, Leung R, Kimokoti R, Bazargan-Hejazi S, Hay SI, Yadgir S, Biryukov S, Vollset SE, Alam T, Frank T, Farid T, Miller T, Vos T, Barnighausen T, Gebrehiwot TT, Yano Y, Al-Aly Z, Mehari A, Handal A, Kandel A, Anderson B, Biroscak B, Mozaffarian D, Dorsey ER, Ding EL, Park EK, Wagner G, Hu G, Chen H, Sunshine JE, Khubchandani J, Leasher J, Leung J, Salomon J, Unutzer J, Cahill L, Cooper L, Horino M, Brauer M, Breitborde N, Hotez P, Topor-Madry R, Soneji S, Stranges S, James S, Amrock S, Jayaraman S, Patel T, Akinyemiju T, Skirbekk V, Kinfu Y, Bhutta Z, Jonas JB, Murray CJL. The State of US Health, 1990-2016: Burden of Diseases, Injuries, and Risk Factors Among US States. JAMA. 2018 Apr 10;319(14):1444-1472. doi: 10.1001/jama.2018.0158. PMID 29634829
- [Result] Steventon A, Bardsley M, Billings J, Dixon J, Doll H, Beynon M, Hirani S, Cartwright M, Rixon L, Knapp M, Henderson C, Rogers A, Hendy J, Fitzpatrick R, Newman S. Effect of telecare on use of health and social care services: findings from the Whole Systems Demonstrator cluster randomised trial. Age Ageing. 2013 Jul;42(4):501-8. doi: 10.1093/ageing/aft008. Epub 2013 Feb 25. PMID 23443509
- [Result] Steventon A, Bardsley M, Billings J, Dixon J, Doll H, Hirani S, Cartwright M, Rixon L, Knapp M, Henderson C, Rogers A, Fitzpatrick R, Hendy J, Newman S; Whole System Demonstrator Evaluation Team. Effect of telehealth on use of secondary care and mortality: findings from the Whole System Demonstrator cluster randomised trial. BMJ. 2012 Jun 21;344:e3874. doi: 10.1136/bmj.e3874. PMID 22723612
- [Result] Hirani SP, Rixon L, Beynon M, Cartwright M, Cleanthous S, Selva A, Sanders C, Newman SP; WSD investigators. Quantifying beliefs regarding telehealth: Development of the Whole Systems Demonstrator Service User Technology Acceptability Questionnaire. J Telemed Telecare. 2017 May;23(4):460-469. doi: 10.1177/1357633X16649531. Epub 2016 May 25. PMID 27224997
- [Result] Steventon A, Grieve R, Bardsley M. An Approach to Assess Generalizability in Comparative Effectiveness Research: A Case Study of the Whole Systems Demonstrator Cluster Randomized Trial Comparing Telehealth with Usual Care for Patients with Chronic Health Conditions. Med Decis Making. 2015 Nov;35(8):1023-36. doi: 10.1177/0272989X15585131. Epub 2015 May 18. PMID 25986472
- [Result] Bardsley M, Steventon A, Doll H. Impact of telehealth on general practice contacts: findings from the whole systems demonstrator cluster randomised trial. BMC Health Serv Res. 2013 Oct 8;13:395. doi: 10.1186/1472-6963-13-395. PMID 24099334
- [Result] Owusu Obeng A, Fei K, Levy KD, Elsey AR, Pollin TI, Ramirez AH, Weitzel KW, Horowitz CR. Physician-Reported Benefits and Barriers to Clinical Implementation of Genomic Medicine: A Multi-Site IGNITE-Network Survey. J Pers Med. 2018 Jul 24;8(3):24. doi: 10.3390/jpm8030024. PMID 30042363
- [Result] Kimura BJ, Shaw DJ, Amundson SA, Phan JN, Blanchard DG, DeMaria AN. Cardiac Limited Ultrasound Examination Techniques to Augment the Bedside Cardiac Physical Examination. J Ultrasound Med. 2015 Sep;34(9):1683-90. doi: 10.7863/ultra.15.14.09002. Epub 2015 Aug 12. PMID 26269293
- [Result] Halcox JPJ, Wareham K, Cardew A, Gilmore M, Barry JP, Phillips C, Gravenor MB. Assessment of Remote Heart Rhythm Sampling Using the AliveCor Heart Monitor to Screen for Atrial Fibrillation: The REHEARSE-AF Study. Circulation. 2017 Nov 7;136(19):1784-1794. doi: 10.1161/CIRCULATIONAHA.117.030583. Epub 2017 Aug 28. PMID 28851729
- [Result] Weinfurt KP, Hernandez AF, Coronado GD, DeBar LL, Dember LM, Green BB, Heagerty PJ, Huang SS, James KT, Jarvik JG, Larson EB, Mor V, Platt R, Rosenthal GE, Septimus EJ, Simon GE, Staman KL, Sugarman J, Vazquez M, Zatzick D, Curtis LH. Pragmatic clinical trials embedded in healthcare systems: generalizable lessons from the NIH Collaboratory. BMC Med Res Methodol. 2017 Sep 18;17(1):144. doi: 10.1186/s12874-017-0420-7. PMID 28923013
- See also: Related Info — https://enews.wvu.edu/articles/2018/10/02/wvu-partners-with-national-heart-group-to-offer-free-exams